CLINICAL TRIAL: NCT06755424
Title: Goat Milk-based Infant Formula and the Prevalence of Gastrointestinal Symptoms in Infants: a Real-world-evidence Study from Brazil, Mexico, Russia, and the Netherlands
Brief Title: GI Symptoms in Infants Fed Goat Milk-based Infant Formula
Status: Completed | Type: Observational
Sponsor: Ausnutria Hyproca B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: P21-013
Record Dates: First submitted 2024-12-17; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Stool Assessment; Skin Rash; Urticaria; Regurgitation; Respiratory Ilness; Crying Time in Colicky Infants; Bloating; DIARRHEA, INFANTILE; Constipation
Keywords: gastrointestinal symptoms; CoMiSS; consumer survey; goat milk-based infant formula
MeSH Terms: conditions — Exanthema; Urticaria; Gastroesophageal Reflux; Diarrhea, Infantile; Constipation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GMF-consumers and GMF-non-consumers: Intervention of interest commercially available Kabrita® stage 1 or 2 compared to any other infant formula type

SUMMARY:
A cross-sectional observational survey was conducted in Brazil, Mexico, Russia, and The Netherlands by recruiting parents/legal guardians through social media. Gastrointestinal symptoms after introduction of Goat milk-based infant formula (GMF) were questioned using the validated Cow's Milk-Related Symptom Score (CoMiSS®; scoring 0-33), lower scores indicate fewer symptoms. Occurrence of crying, gassiness, eczema, respiratory symptoms and stool consistency were asked retrospectively before and ≥14 days after introduction of GMF.

DETAILED DESCRIPTION:
A cross-sectional observational online anonymous survey on GI symptoms in infants aged 0-24 months fed GMF has been developed and conducted in Brazil, Mexico, Russia, and The Netherlands. The GMF of interest was commercially available Kabrita® stage 1 or 2 (Ausnutria, B.V., the Netherlands). Participants who had purchased Kabrita® were asked to complete a voluntary survey regarding their experience and observation on their infant's GI complaints. No inclusion criteria were set at the time point of sending out the survey. The survey consisted of 30 questions and was online from June 2021 until November 2022. The survey and associated data collection do not meet the criteria for human subject research and therefore approval by an institutional and/or licensing committee is not needed, and participant consent is not required. Participation in the survey was anonymized and completely voluntary.

ELIGIBILITY:
Inclusion Criteria:

* infants aged 0-24 months
* fed at least once with goat milk-based infants formula

Exclusion Criteria:

* infants aged >24 months
* taking medication for functional GI disorders

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infants aged 0-24 months
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
GI symptoms as assessed by the Cow's Milk-Related Symptom Score (CoMiSS®) after introduction of GMF | 14 days
  Cow's Milk-Related Symptom Score (CoMiSS®; scoring 0-33), lower scores indicate fewer symptoms. The CoMiSS® was developed by an expert panel to increase the awareness of health care professionals for the presence and severity of symptoms, which might be related to cow's milk protein intake. The CoMiSS® is a validated and easy-to-use clinical tool with an estimated sensitivity between 20-77% and a specificity of 54-92% to suspected cow's milk allergy. The CoMiSS® assesses the stool pattern using the Bristol Scale (hard stools, normal stools, soft stools, liquid stools, watery stools); skin symptoms of atopic eczema on head, neck and/or trunk as well as on arms, hands and/or feet; skin symptoms of urticaria; respiratory symptoms, regurgitation; and crying without any obvious cause in hours per day. The total score ranges from 0-33, where lower scores indicate less severe symptoms

SECONDARY OUTCOMES:
retrospective assessment GI symptoms before introduction of Kabrita® and improvement minimally 14 days after introduction. | 14 days
  The survey inquired about GI symptoms before and after introduction of GMF (no score on a scale). These symptoms included gassiness (specified as burping, passing gas, bloating, abdominal pain and/or colic); skin symptoms (specified as rashes, and/or eczema); watery stools/diarrhoea; hard stools/constipation; crying without any obvious cause.
  Questions before switching to GMF: minor GI complaints (y/n). If yes, which complaints (choices: Gassiness / Skin symptoms / Watery stools/diarrhoea / Hard stools/constipation / None). Tendency to cry without any obvious cause (y/n) Questions after switching to GMF: experienced less complaints (y/n). If yes, which complaints improved (choices: Gassiness / Skin symptoms / Watery stools/diarrhoea / Hard stools/constipation / None of the above). Tendency to cry without any obvious cause (choices: Yes, similar as before / Yes, less than before / Yes, worse than before / No). Crying: on average each day (choices: <1, 1-1.5, 1.5-2, 2-3, 3-4, 4-5, >5h)

CONTACTS AND LOCATIONS:
Locations (1):
- Ausnutria B.V, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knipping K, Bohme J, Goossens D, van Lee L, van der Zee L. Goat Milk-Based Infant Formula and the Prevalence of Gastrointestinal Symptoms in Infants: A Real-World-Evidence Study From Brazil, Mexico, Russia, and the Netherlands. Health Sci Rep. 2025 Feb 10;8(2):e70448. doi: 10.1002/hsr2.70448. eCollection 2025 Feb. PMID 39935845